CLINICAL TRIAL: NCT04567953
Title: COVID-19 Tests With Saliva Specimens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Paradigm Laboratories LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PLRD202001
Record Dates: First submitted 2020-09-25; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Saliva and NP paired specimen collection (Experimental)
  Interventions: Other: Saliva collection

INTERVENTIONS:
Other: Saliva collection — Use Spectrum Solutions SDNA1000 or Orasure collection kit or dry tube to collect 1-3 ml of saliva

SUMMARY:
Upper respiratory swabs, such as the nasopharyngeal (NP) swab, have so far been major specimen sources used for the SARS-COV-2 molecular test. However, due to the discomfort and invasiveness of NP collection, and the expense of personal protective equipment, alternative sampling sources such as saliva are desired. The purpose of this proposed study is: 1) to examine whether saliva can be used as an specimen for the SARS-COV-2 molecular test; 2) to test if gingival crevicular fluids is a reliable specimen for the SARS-COV-2 antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Persons referred for COVID-19 testing including those with COVID-19 symptoms and/or a suspected SARS-COV-2 infection or undergoing surveillance testing and

  * Is able to give informed consent
  * Is able to understand oral or written instructions, and
  * Is able to mentally and physically perform self-collection of saliva using the provided collection device.

Exclusion Criteria:

* - Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Employees of Paradigm lab and the assisted living facilities involved in the study
* Members of other vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-06-27 (Estimated)

PRIMARY OUTCOMES:
The clinical evaluation of saliva as specimen for COVID-19 molecular test | 1 hour
  We will evaluate the positive and negative agreement of saliva with nasopharyngeal swab as specimens for COVID-19 molecular test.

CONTACTS AND LOCATIONS:
Overall Officials: Wenli Zhou, PhD, Principal Investigator — Paradigm Laboratories
Locations (1):
- Paradigm Laboratories, Tucson, Arizona, United States